CLINICAL TRIAL: NCT04534036
Title: A 12-week Randomized, Double-Blind Controlled Trial to Evaluate the Tolerability and Gastrointestinal Response of a Novel, Multi-Strain Synbiotic (PDS-08™) in Children Ages 3-17
Brief Title: Tolerability and Functional Assessment of a Novel Children's Synbiotic
Acronym: PDS-08™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seed Health (Industry)
Collaborators: Curebase Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDS-08
Record Dates: First submitted 2020-08-25; First posted 2020-09-01 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Constipation; Signs and Symptoms; Digestive Signs and Symptoms; Infrequent or Difficult Evacuation
MeSH Terms: conditions — Constipation; Signs and Symptoms; Signs and Symptoms, Digestive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Strain Synbiotic (PDS-08) (Active Comparator): PDS-08 is a rationally defined microbial consortium consisting of 9 strains, with FOS-inulin as prebiotic. Participants will be instructed to take 1 sachet daily for the duration of the trial.
  Interventions: Dietary Supplement: PDS-08
- Placebo (Placebo Comparator): Placebo sachets for PDS-08 will contain potato or tapioca maltodextrin matched for color and texture. Participants will be instructed to take 1 sachet daily for the duration of the trial.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: PDS-08 — PDS-08 is a novel synbiotic comprised of nine probiotic bacterial strains and FOS-inulin as a prebiotic.
  Arms: Multi-Strain Synbiotic (PDS-08)
Other: Placebo — Placebo sachets will contain potato or tapioca maltodextrin.
  Arms: Placebo

SUMMARY:
Recent data support the use of specific probiotic strains in a pediatric population. However, given the wide number of commercial products available, and contradictory data in the literature, healthcare providers and consumers are uncertain about whether or not to use probiotics in children and which one(s) to choose. While much progress has been made in understanding the gastrointestinal microbiota and its role in the balanced development of the infant immune system, the tolerability and efficacy of introducing beneficial microbes into the pediatric gastrointestinal tract remain underexplored.

The purpose of this study is to investigate the effect of a 9 strain synbiotic consortium comprised of strains with previous pediatric clinical data for use in modulating airway sensitivity, gastrointestinal discomfort, dermatological inflammation, and reduction in the duration and severity of upper respiratory tract infections in a pediatric population.

DETAILED DESCRIPTION:
During infancy and childhood, environmental factors including the maternal vaginal and skin microbiomes, breast milk microbiota, breast milk, geographic location, and use of antibiotics will exert significant influence over the offspring's microbiota and have a determinant impact on their health later in life. Unfavorable environmental exposures, coupled with an immature immune system in early life can, therefore, confer suboptimal immune responses that can lead to the development of extra-gastrointestinal conditions such as allergic rhinitis, asthma, and atopic dermatitis-which affects 15-20% of the world's population. Furthermore, while the indiscriminate use of antibiotics has decreased, they remain standard-of-care for most childhood infections, and unfortunately, often result in short- or long-term disruption of the patient's microbiome.

Constipation is a common childhood gastrointestinal disorder, with a worldwide prevalence between 0.7-29.6%. Its etiology is multifactorial and usually not due to underlying conditions. Few studies have explored the implications of the intestinal or fecal microbiota in childhood constipation, yet some have shown benefits of various probiotic compositions in reducing transit time and improving bowel movement frequency. Dysbiosis of the gut microbiome may play an important role in functional constipation.

PDS-08™ is a novel synbiotic, comprised of nine probiotic bacterial strains and fructooligosaccharide with inulin (FOS-inulin) as a prebiotic. A synbiotic is defined as a probiotic ("live microorganisms that, when administered in adequate amounts, confer a health benefit on the host") plus an established prebiotic ("a substrate that is selectively utilized by host microorganisms conferring a health benefit")-or, an untested live microbe co-administered with a substrate that it selectively utilizes. The selected probiotics and prebiotic in the PDS-08 formulation have shown to improve antibiotic-associated diarrhea, gastrointestinal and respiratory tract infections, allergic rhinitis, atopic dermatitis, irritable bowel syndrome (IBS) symptoms, and/or microbiota modulation. The positive outcomes of these respective studies warrants further investigation of the strains as part of a probiotic consortium with the potential to modulate the microbiota, regulate dysbiosis, and confer a benefit to host health. There is a need for additional systematic studies on probiotic administration in pediatric populations, with a focus on measuring shifts in the fecal microbiota and markers of gut health and function. Therefore, the objective of this study is to assess the efficacy, tolerability, and safety of a novel synbiotic in healthy children with occasional constipation, over 12 weeks, as compared to a sensory-matched placebo.

This is a randomized, 12-week study to compare the efficacy and tolerability of PDS-08 in a cohort of 100 healthy children with constipation. 50 subjects will receive PDS-08™ over 12 weeks, and 50 subjects will receive a placebo. Subjects will provide stool samples at baseline and week 12. Safety is a paramount concern in the study design and will be monitored carefully throughout the study. Parents or direct relative guardians of study subjects will receive extensive education on synbiotic use.

ELIGIBILITY:
Inclusion Criteria:

* The parent(s) or direct relative guardian(s) of the participant must be willing and able to give informed assent/consent for participation in the study.
* Participant must be in good health as determined from participant's medical history.
* Males & Females between 3-17 years old.
* Normal weight or overweight (BMI between the age- and sex-specific 5th percentile and 95th percentile).
* Children with constipation (defined as less than 4 bowel movements per week) and/or baseline Bristol Stool Form Scale score of 1 or 2.
* Participant's parent(s) must be willing and able (in the PI's opinion) to comply with all study requirements.
* Children with healthy skin or eczema and/or acne.
* Females of childbearing potential (post-menarche) and/or their parents must make a written and/or verbal statement prior to randomization indicating that they are not pregnant and adhere to a pregnancy prevention method (abstinence or barrier method plus spermicidal foam or oral or implanted contraceptive).
* Consistent use of medications not listed in the exclusion criteria.
* Participant is under the care of a parent or direct relative guardian.

Exclusion Criteria:

* Underweight (BMI<5th percentile for age) or obese (BMI above the 95th percentile on the Centers for Disease Control and Prevention growth charts).
* Participants are taking, and plan to continue taking, medications (including over the counter (OTC), such as simethicone for gas), home remedies (such as juice for constipation), herbal preparations, or rehydration fluids that might affect GI tolerance.
* Participants taking laxatives.
* Participants using probiotics, antibiotics, or antifungals during the course of the study or within the past 1 month.
* Participants receiving administration of any investigational drug within the past 1 month.
* Participants who are pregnant, lactating, or planning a pregnancy during the course of the study.
* Participants with compromised immunity.
* Participants with GI disease (e.g., inflammatory bowel disease, celiac disease, prior intestinal resection, SIBO/small intestinal bacterial growth, irritable bowel syndrome, functional abdominal pain, or lactose intolerance).
* Participants are taking medication such as antipsychotics, antidepressants, mood stabilizers, medications for Attention Deficit Hyperactivity Disorder, anti-anxiety medications (Anxiolytics), or related medication.
* Participants on medically prescribed diets or supplements other than a standard multivitamin.
* Participants with plans to travel outside the USA during the study. Alcohol or drug abuse.
* Participants using any oral over the counter or prescription medications for acne or atopic dermatitis.
* Participants who have recently tested positive for COVID-19 or who live with adults with an active COVID-19 infection.
* Participants are under the care of someone other than a parent or direct relative guardian.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who are spontaneous bowel movement responders, defined as having an average of ≥ 4 complete spontaneous bowel movements (CSBMs) per week and an average increase of ≥ 1 CSBM from baseline, by age group: 3-6, 7-12, 13-17 years. | Baseline-Day 84
  Assessed as the change from baseline and compared to placebo for the continuous variable estimated using a linear mixed model.

SECONDARY OUTCOMES:
Average increase from baseline of Bristol Stool Form Scale (BSFS) score by ≥ 1 point (stool characterized as an increase to either type 2 or 3 or 4) in the intervention group, compared to the placebo group. | Baseline-Day 84
  Assessed by daily stool characteristics reported using the seven-point ordinal BSFS score. The BSFS classifies human stool into seven types and scores them accordingly. Type 1: Separate hard lumps (hard to pass) Type 2: Sausage-shaped and lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage, smooth and soft Type 5: Soft blobs with clear cut edges (passed easily) Type 6: Fluffy pieces with ragged edges, a mushy stool Type 7: Watery, no solid pieces, entirely liquid. Types 1 and 2 indicate constipation, with 3 through 5 represent the ideal stool form, and 6 and 7 tend towards diarrhea.
  For a given assessment week, the weekly stool consistency is defined as the sum of non-missing stool consistency score for spontaneous bowel movements during that week divided by the number of non-missing stool consistency scores for spontaneous bowel movements during that week. The parameter will be analyzed using a linear mixed model.
Decrease of ≥ 10% in time spent emptying bowel from beginning to end of bowel movement, compared to baseline. | Baseline-Day 84
Changes in subjective assessment of gut tolerability as reported by parents or direct relative guardians, indicated by sustained (longer than 7 days of) abdominal pain, severe bloating, heartburn, acid reflux, or indigestion. | Baseline-Day 84
  Assessed by online daily symptom-tracking of stool-quality, regularity, ease of expulsion, bloating, and flatulence.
Maintenance or increase of diversity within the PDS-08 treatment group. | Baseline-Day 84
  Microbiota composition will be identified through fecal samples for total genomic DNA extraction in participants supplemented with PDS-08 or placebo. Metagenomic sequencing will yield a total observable species count and maintenance will be defined as within 20% of the total observed species count when compared to baseline.
Significant increase in QoL measured by the KINDL questionnaire with respect to mean change from baseline score (p<0.05). | Baseline-Day 84
Exploratory: number of respiratory tract infections in the PDS-08 group compared to placebo. | Baseline-Day 84
Exploratory: number and percent of participants with reduction in number of acne lesions from baseline as measured by global count of blemishes. | Baseline-Day 84
Exploratory outcomes: changes in fecal calprotectin, histamine, bacterial enzymes (β-glucosidase and β-glucuronidase), β-defensin (hBD2) and short chain fatty acids in treatment group compared to the placebo group. | Baseline-Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Charles Baum, MD, Principal Investigator — Encore Health
Locations (1):
- Curebase, Inc., San Francisco, California, United States

REFERENCES:
- [Background] Candela M, Biagi E, Maccaferri S, Turroni S, Brigidi P. Intestinal microbiota is a plastic factor responding to environmental changes. Trends Microbiol. 2012 Aug;20(8):385-91. doi: 10.1016/j.tim.2012.05.003. Epub 2012 Jun 5. PMID 22672911
- [Background] Jost T, Lacroix C, Braegger C, Chassard C. Assessment of bacterial diversity in breast milk using culture-dependent and culture-independent approaches. Br J Nutr. 2013 Oct;110(7):1253-62. doi: 10.1017/S0007114513000597. Epub 2013 Mar 14. PMID 23507238
- [Background] Morrow AL, Ruiz-Palacios GM, Altaye M, Jiang X, Guerrero ML, Meinzen-Derr JK, Farkas T, Chaturvedi P, Pickering LK, Newburg DS. Human milk oligosaccharides are associated with protection against diarrhea in breast-fed infants. J Pediatr. 2004 Sep;145(3):297-303. doi: 10.1016/j.jpeds.2004.04.054. PMID 15343178
- [Background] Schuez-Havupalo L, Toivonen L, Karppinen S, Kaljonen A, Peltola V. Daycare attendance and respiratory tract infections: a prospective birth cohort study. BMJ Open. 2017 Sep 5;7(9):e014635. doi: 10.1136/bmjopen-2016-014635. PMID 28877939
- [Background] Ngurah G, Putra S, Suraatmaja S, Ketut I, Aryasa N. Effect of probiotics supplementation on acute diarrhea in infants: a randomized double blind clinical trial. Paediatrica Indonesiana. 2007;47.
- [Background] Ege MJ, Mayer M, Normand AC, Genuneit J, Cookson WO, Braun-Fahrlander C, Heederik D, Piarroux R, von Mutius E; GABRIELA Transregio 22 Study Group. Exposure to environmental microorganisms and childhood asthma. N Engl J Med. 2011 Feb 24;364(8):701-9. doi: 10.1056/NEJMoa1007302. PMID 21345099
- [Background] Avena-Woods C. Overview of atopic dermatitis. Am J Manag Care. 2017 Jun;23(8 Suppl):S115-S123. PMID 28978208
- [Background] Gensollen T, Blumberg RS. Correlation between early-life regulation of the immune system by microbiota and allergy development. J Allergy Clin Immunol. 2017 Apr;139(4):1084-1091. doi: 10.1016/j.jaci.2017.02.011. PMID 28390575
- [Background] Vaz LE, Kleinman KP, Raebel MA, Nordin JD, Lakoma MD, Dutta-Linn MM, Finkelstein JA. Recent trends in outpatient antibiotic use in children. Pediatrics. 2014 Mar;133(3):375-85. doi: 10.1542/peds.2013-2903. Epub 2014 Feb 2. PMID 24488744
- [Background] Wistrom J, Norrby SR, Myhre EB, Eriksson S, Granstrom G, Lagergren L, Englund G, Nord CE, Svenungsson B. Frequency of antibiotic-associated diarrhoea in 2462 antibiotic-treated hospitalized patients: a prospective study. J Antimicrob Chemother. 2001 Jan;47(1):43-50. doi: 10.1093/jac/47.1.43. PMID 11152430
- [Background] van den Berg MM, Benninga MA, Di Lorenzo C. Epidemiology of childhood constipation: a systematic review. Am J Gastroenterol. 2006 Oct;101(10):2401-9. doi: 10.1111/j.1572-0241.2006.00771.x. PMID 17032205
- [Background] Sadeghzadeh M, Rabieefar A, Khoshnevisasl P, Mousavinasab N, Eftekhari K. The effect of probiotics on childhood constipation: a randomized controlled double blind clinical trial. Int J Pediatr. 2014;2014:937212. doi: 10.1155/2014/937212. Epub 2014 Apr 9. PMID 24812563
- [Background] Bu LN, Chang MH, Ni YH, Chen HL, Cheng CC. Lactobacillus casei rhamnosus Lcr35 in children with chronic constipation. Pediatr Int. 2007 Aug;49(4):485-90. doi: 10.1111/j.1442-200X.2007.02397.x. PMID 17587273
- [Background] de Meij TG, de Groot EF, Eck A, Budding AE, Kneepkens CM, Benninga MA, van Bodegraven AA, Savelkoul PH. Characterization of Microbiota in Children with Chronic Functional Constipation. PLoS One. 2016 Oct 19;11(10):e0164731. doi: 10.1371/journal.pone.0164731. eCollection 2016. PMID 27760208
- [Background] Zhu L, Liu W, Alkhouri R, Baker RD, Bard JE, Quigley EM, Baker SS. Structural changes in the gut microbiome of constipated patients. Physiol Genomics. 2014 Sep 15;46(18):679-86. doi: 10.1152/physiolgenomics.00082.2014. Epub 2014 Jul 29. PMID 25073603
- [Background] Zoppi G, Cinquetti M, Luciano A, Benini A, Muner A, Bertazzoni Minelli E. The intestinal ecosystem in chronic functional constipation. Acta Paediatr. 1998 Aug;87(8):836-41. doi: 10.1080/080352598750013590. PMID 9736230
- [Background] de Souza Lima Sant'Anna M, Rodrigues VC, Araujo TF, de Oliveira TT, do Carmo Gouveia Peluzio M, de Luces Fortes Ferreira CL. Yacon-Based Product in the Modulation of Intestinal Constipation. J Med Food. 2015 Sep;18(9):980-6. doi: 10.1089/jmf.2014.0115. Epub 2015 Feb 18. PMID 25692980
- [Background] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Background] Swanson KS, Gibson GR, Hutkins R, Reimer RA, Reid G, Verbeke K, Scott KP, Holscher HD, Azad MB, Delzenne NM, Sanders ME. The International Scientific Association for Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of synbiotics. Nat Rev Gastroenterol Hepatol. 2020 Nov;17(11):687-701. doi: 10.1038/s41575-020-0344-2. Epub 2020 Aug 21. PMID 32826966
- [Background] Gibson GR, Hutkins R, Sanders ME, Prescott SL, Reimer RA, Salminen SJ, Scott K, Stanton C, Swanson KS, Cani PD, Verbeke K, Reid G. Expert consensus document: The International Scientific Association for Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of prebiotics. Nat Rev Gastroenterol Hepatol. 2017 Aug;14(8):491-502. doi: 10.1038/nrgastro.2017.75. Epub 2017 Jun 14. PMID 28611480
- [Background] Shornikova AV, Casas IA, Isolauri E, Mykkanen H, Vesikari T. Lactobacillus reuteri as a therapeutic agent in acute diarrhea in young children. J Pediatr Gastroenterol Nutr. 1997 Apr;24(4):399-404. doi: 10.1097/00005176-199704000-00008. PMID 9144122
- [Background] Shornikova AV, Casas IA, Mykkanen H, Salo E, Vesikari T. Bacteriotherapy with Lactobacillus reuteri in rotavirus gastroenteritis. Pediatr Infect Dis J. 1997 Dec;16(12):1103-7. doi: 10.1097/00006454-199712000-00002. PMID 9427453
- [Background] Quigley EM. The efficacy of probiotics in IBS. J Clin Gastroenterol. 2008 Jul;42 Suppl 2:S85-90. doi: 10.1097/MCG.0b013e31816244ca. PMID 18542036